CLINICAL TRIAL: NCT07370961
Title: CKD-aP: Diagnosis and Treatment Through a Multidisciplinary Approach - Pilot Study
Brief Title: Pilot Study to Evaluate the Impact of a Multidisciplinary Approach (Pharmacological and Psychological) in the Treatment of Chronic Kidney Disease-Associated Pruritus
Acronym: CKD-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Federico Alberici, Prof., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NP 6183
Record Dates: First submitted 2025-12-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease-associated Pruritus
Keywords: Chronic Kidney Disease-associated Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): standard of care alone
- Intervention (Experimental): standard of care plus a structured psychological intervention
  Interventions: Other: Structured psychological intervention

INTERVENTIONS:
Other: Structured psychological intervention — Structured psychological intervention
  Arms: Intervention

SUMMARY:
This is a single-center, pilot, randomized, open-label, non-profit interventional study designed to evaluate the impact of a multidisciplinary approach on chronic kidney disease-associated pruritus (CKD-aP) in patients undergoing chronic extracorporeal hemodialysis.

Twenty adult, clinically stable hemodialysis patients with moderate to severe uremic pruritus will be enrolled and randomized to receive either standard of care alone or standard of care plus a structured psychological intervention. The primary objective is to assess the change in pruritus-related quality of life after 6 months, measured by the KDQOL-SF questionnaire. Secondary objectives include evaluation of pruritus severity, quality of life, sleep quality, psychological distress, patient engagement, clinical and biochemical parameters, and exploration of patients' psychological experience over time.

The study aims to provide preliminary evidence on the effectiveness of integrating psychological support into the management of CKD-associated pruritus in the hemodialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* KDQOL-SF™ 1.3 score ≥ 3 (corresponding to the presence of the symptom in the last 4 weeks, rated as "moderately bothered")
* On chronic hemodialysis for at least 3 months and clinically stable
* Signed informed consent for participation in the study

Exclusion Criteria:

* Refusal to provide informed consent
* Age < 18 years
* KDQOL-SF™ 1.3 score < 3
* Pruritus secondary to dermatologic diseases, autoimmune diseases with skin involvement (e.g. SLE, scleroderma, vasculitis, etc.), hepatobiliary diseases causing cholestatic jaundice, malignancies, or uncontrolled endocrine disorders
* Active substance abuse
* Severe mental illness or severe cognitive impairment (e.g. active psychosis, dementia, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 months in the pruritus intensity-related item of the Kidney Disease Quality of Life - Short Form (KDQOL-SF) questionnaire. | 6 months
  Change from baseline to 6 months in the pruritus intensity-related item of the Kidney Disease Quality of Life - Short Form (KDQOL-SF) questionnaire. This item assesses how bothersome pruritus is, on a scale ranging from 1 (not bothered at all) to 5 (extremely bothered).

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Italy, Italy

IPD SHARING:
Plan to Share IPD: No